CLINICAL TRIAL: NCT01005407
Title: An Observer-Blinded, Randomized, Parallel-Group, Multi-Center Study Comparing the Safety and Immunogenicity of HEPLISAV™ to Licensed Vaccine (Engerix-B®) Among Healthy Subjects 40 to 70 Years of Age
Brief Title: Safety and Immunogenicity Study of the Hepatitis B Virus (HBV) Vaccine, HEPLISAV Compared to Engerix-B Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DV2-HBV-16
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Results first posted 2018-01-11 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: HBV vaccine; Hepatitis B vaccine; Hepatitis B; Hepatitis; HBV; Prevention & Control; Healthy; Healthy volunteers
MeSH Terms: conditions — Hepatitis B; Hepatitis | interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HEPLISAV and/or Placebo (Experimental): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018)
  Interventions: Biological: HEPLISAV and/or Placebo
- Engerix-B(1) (Active Comparator): 1.0 mL Engerix-B
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: HEPLISAV and/or Placebo — Intramuscular (IM) injections on Week 0 and Week 4; placebo (saline) injection at Week 24
  Other Names: Hepatitis B vaccine (recombinant), adjuvanted
  Arms: HEPLISAV and/or Placebo
Biological: Engerix-B — Intramuscular (IM) injections on Week 0, Week 4 and Week 24
  Other Names: Hepatitis B vaccine (recombinant)
  Arms: Engerix-B(1)

SUMMARY:
The purpose of the study is to evaluate the safety, immunogenicity and lot-to-lot consistency of an investigational hepatitis B virus vaccine, HEPLISAV™, in healthy adults 40 to 70 years of age

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety, immunogenicity and lot-to-lot consistency of an investigational hepatitis B virus vaccine, HEPLISAV™, in healthy adults 40 to 70 years of age

ELIGIBILITY:
Inclusion Criteria:

* be 40 - 70 years of age, inclusive
* be seronegative for hepatitis B surface antigen (HBsAg), antibody against hepatitis B surface antigen (anti-HBsAg), antibody against hepatitis B core antigen (anti-HBcAg), and human immunodeficiency virus (HIV)
* be in good health in the opinion of the investigator, based upon medical history, physical examination, and laboratory evaluation
* if female of childbearing potential, agree to consistently use a highly effective method of birth control from screening visit through the treatment phase, for up to 28 days after the last injection

Exclusion Criteria:

* if female of childbearing potential, is pregnant, breastfeeding, or planning a pregnancy
* has a history of or is considered by the investigator to be at high risk for recent exposure to HBV or HIV; for example, current intravenous drug use or has unprotected sex with known HBV/HIV positive partner
* has a known history of autoimmune disease
* has previously received any hepatitis B vaccine (approved or investigational)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2452 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (29):
  - Huntsville, Alabama
  - San Diego, California
  - Santa Ana, California
  - Denver, Colorado
  - Melbourne, Florida
  - Pinellas Park, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - South Bend, Indiana
  - Rockville, Maryland
  - Brooklyn Center, Minnesota
  - Edina, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Rochester, New York
  - Cincinnati, Ohio
  - Erie, Pennsylvania
  - Grove City, Pennsylvania
  - Jefferson Hills, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Upper Saint Clair, Pennsylvania
  - Anderson, South Carolina
  - Greer, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Canada (3):
  - Mount Pearl, Newfoundland and Labrador
  - Toronto, Ontario
  - Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heyward WL, Kyle M, Blumenau J, Davis M, Reisinger K, Kabongo ML, Bennett S, Janssen RS, Namini H, Martin JT. Immunogenicity and safety of an investigational hepatitis B vaccine with a Toll-like receptor 9 agonist adjuvant (HBsAg-1018) compared to a licensed hepatitis B vaccine in healthy adults 40-70 years of age. Vaccine. 2013 Nov 4;31(46):5300-5. doi: 10.1016/j.vaccine.2013.05.068. Epub 2013 May 30. PMID 23727002

RESULTS

PARTICIPANT FLOW:
Groups:
- HEPLISAV and/or Placebo: 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018)
  HEPLISAV and/or Placebo: Intramuscular (IM) injections at Week 0, Week 4, plus a placebo (saline) injection at Week 24
- Engerix-B: 1.0 mL Engerix-B
  Engerix-B: Intramuscular injections at Week 0, Week 4, and Week 24
Period: Overall Study
Arm/Group | HEPLISAV and/or Placebo | Engerix-B
Started | 1969 | 483
Completed | 1818 | 451
Not Completed | 151 | 32

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 study injection and who had any post-baseline safety data
Groups:
- HEPLISAV and Placebo: 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018)
  HEPLISAV and/or Placebo: Intramuscular (IM) injections at Week 0, Week 4, plus a placebo (saline) injection at Week 24
- Engerix-B: 1.0 mL Engerix-B
  Engerix-B: Intramuscular (IM) injections on Week 0, Week 4 and Week 24
- Total: Total of all reporting groups
Arm/Group | HEPLISAV and Placebo | Engerix-B | Total
Number analyzed (Participants) | 1968 | 481 | 2449
Age, Customized [Count of Participants; unit: Participants]
  ≥ 40 to ≤ 70 years | 1968 | 481 | 2449
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1025 | 245 | 1270
  Male | 943 | 236 | 1179
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 151 | 45 | 196
  United States | 1817 | 436 | 2253

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Have a Seroprotective Immune Response
Description: Percentage of subjects who have a seroprotective immune response (anti-HBsAg antibody≥ 10 milli-international unit (mIU)/mL) 8 weeks after the last active dose of HEPLISAV™ compared to 8 weeks after the last active dose of Engerix-B®
Time Frame: at Week 12 and at Week 32
Population: Non-Inferiority per Protocol population:Randomized subjects who received 1 of 3 consistency lots of HEPLISAV or Engerix-B within the study visit windows, had all 3 study injections as randomized and within the study visit windows, no major protocol deviations, and anti-HBs levels obtained within study visit windows at baseline, Week 12, and Week 32
Measure: Number; unit: Percentage of participants
Arm/Group | HEPLISAV and Placebo | Engerix-B
Number analyzed (Participants) | 1121 | 353
Percentage of participants | 90.1 | 70.5

2. Secondary Outcome: Percentage of Participants With Local and Systemic Reaction to Injections
Time Frame: within 7 days for post-injection reactions
Population: Safety population: All participants who received at least 1 study injection and had at least 1 post-baseline safety data. NOTE: Only subjects with non-missing injection results in the Safety population are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | HEPLISAV and Placebo | Engerix-B
Number analyzed (Participants) | 1952 | 477
percentage of participants
  Local reaction: Injection 1 | 24.33 | 18.87
  Local reaction: Injection 2 | 23.10 | 16.16
  Local reaction: Injection 3 | 0 | 13.84
  Systemic reaction: Injection 1 | 22.34 | 22.64
  Systemic reaction: Injection 2 | 16.38 | 18.10
  Systemic reaction: Injection 3 | 0 | 13.39

ADVERSE EVENTS:
Description: Adverse events were assessed for the safety analysis population: All participants who received at least 1 study injection and had a least 1 post baseline safety data
Arm/Group | HEPLISAV and/or Placebo | Engerix-B(1)
Serious Adverse Events (participants affected / at risk) | 78/1968 | 23/481
Other Adverse Events (participants affected / at risk) | 80/1968 | 25/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV and/or Placebo (N=1968) | Engerix-B(1) (N=481)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cavernous sinus thrombosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Water intoxication (Metabolism and nutrition disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign intracranial hypertension (Nervous system disorders) | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV and/or Placebo (N=1968) | Engerix-B(1) (N=481)
Nasopharyngitis (Infections and infestations) | 80 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less